CLINICAL TRIAL: NCT04575311
Title: A Double-Blind, Randomized, Placebo-Controlled, Single Ascending Dose Study to Investigate the Pharmacokinetic Profile of Oral AB680 in Healthy Volunteers
Brief Title: A Study to Investigate the Pharmacokinetic Profile of Oral AB680 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ARC-11
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — quemliclustat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active: Dose Escalation (Active Comparator): Participants will receive a single oral dose of AB680 at one of two ascending dose levels. Assignment to receive AB680 will be random.
  Interventions: Drug: AB680
- Placebo: Dose Escalation (Placebo Comparator): Participants will receive matching placebo as a single oral dose. Assignment to receive matching placebo will be random.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AB680 — AB680 is a Cluster of Differentiation (CD)73 Inhibitor
  Arms: Active: Dose Escalation
Other: Placebo — Matching Placebo
  Arms: Placebo: Dose Escalation

SUMMARY:
A Double-Blind, Randomized, Placebo-Controlled, Single Ascending Dose Study to Investigate the Pharmacokinetic Profile of Oral AB680 in Healthy Volunteers.

DETAILED DESCRIPTION:
The study will evaluate minimum of 2 dose levels of AB680 in 8 participants per cohort. Cohorts will be gender-balanced to the extent possible, and will be randomized 3:1, active vs placebo, respectively.

The participants will be closely observed for the first 48 hours following drug administration to monitor the general tolerability of AB680.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 55 years, inclusive, at screening
* Body mass index 18 to 32 kilograms/m^2 inclusive
* Willing and able to sign informed consent
* Negative tests for hepatitis B surface antigen, anti-hepatitis C virus, and human immunodeficiency virus (HIV)-1 and HIV-2 antibody at screening
* Healthy as determined by pre-study screening

Exclusion Criteria:

* History of clinically significant drug and/or food allergies
* Positive drug and alcohol screen at screening and (each) admission to the clinical research center.
* Participation in a drug study within 60 days prior to (the first) drug administration in the current study. Participation in more than 4 other drug studies in the 12 months prior to (the first) drug administration in the current study
* Participants who have significant infection or known inflammatory process on screening or admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
AB680 Peak Plasma Concentration (Cmax) | Pre-dose; from First Dose Date to 15 Days After the Last Dose of AB680
  Cmax as measured by the Area Under Concentration-Time Curve from Plasma Collection and Analysis.
AB680 Time of Peak Concentration (Tmax) | Pre-dose; from First Dose Date to 15 Days After the Last Dose of AB680
  Tmax as measured by the Time to Maximum Concentration-Time Curve from Plasma Collection and Analysis
Area under the plasma concentration-time curve from time zero to t hours (AUC 0-t) of AB680 | Pre-dose; from First Dose Date to 15 Days After the Last Dose of AB680

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | From First Dose Date to 15 Days After the Last Dose of AB680
  Number of participants with TEAEs as assessed by CTCAE v5.0.

OTHER OUTCOMES:
Pharmacodynamic (PD) Effects of AB680 | Pre-dose; from First Dose Date to 15 Days After the Last Dose of AB680]
  Enzymatic Activity of CD73 measured in participant blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-11 - Lay Summary (English Version) — https://trials.arcusbio.com/study/?id=ARC-11